CLINICAL TRIAL: NCT01109732
Title: Physical Activity, Function and Quality of Life in Patients After Endovascular Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Oslo University College (Other)
Responsible Party: Principal Investigator, Elisabeth Bø, MSc, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/2192-1
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Systematic physical training (Experimental): Hospital-based SET two days per week for 12 weeks and one home-based exercise session every week. The group-based SET was based on The Norwegian Ullevaal Model, a modified cardiac rehabilitation program, and was slightly adjusted to be applicable to this patient group. Each SET session lasted for 60 minutes and consisted of warm-up exercises, three high-intensity, two moderate-intensity and cool-down exercises, including stretching. The exercises were generally simple aerobic dance movements and walking and involved the use of both upper and lower extremities. The warm-up exercises included large muscle movements that were repeated later in the higher-intensity intervals, but with greater force and a larger range of movement.
  Interventions: Other: Systematic physical training with instructor
- Treatment as of today (No Intervention): The control group did not receive any additional follow-up regarding exercise at discharge beyond the general advice about the importance of exercise that is routinely provided at the hospital.

INTERVENTIONS:
Other: Systematic physical training with instructor — Training 3 times per week for 6 months, the first 3 months with an instructor
  Arms: Systematic physical training

SUMMARY:
The purpose of this study is to investigate how systematic physical training after endovascular treatment influence the durability of the endovascular treatment and how it effects physical function, quality of life and future cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* 55 years old or older
* successful endovascular
* living in Oslo or in the close area being able to come to physical training classes at the hospital

Exclusion Criteria:

* endovascular treatment on study-leg last 2 years
* other reasons for reduced walking function than peripheral arterial disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Time to potential occlusion | 1 year

SECONDARY OUTCOMES:
6 Minutes Walk Test | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Bergland, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No